CLINICAL TRIAL: NCT02464644
Title: A Questionnaire Study on Hereditary Hemorrhagic Telangiectasia (HHT) and Other Medical Conditions, Compared to the General Population
Brief Title: Frequency of Common Medical Conditions in People With and Without HHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CLS/2012/2
Record Dates: First submitted 2012-04-30; First posted 2015-06-08 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Hereditary Hemorrhagic Telangiectasia (HHT)
Keywords: On-line Questionnaire; No travel; Health; Medicines; Drugs; Lifestyle; Family; Help for others; Rare condition; General population
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic | interventions — Surveys and Questionnaires; Confidentiality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- People with HHT (Experimental): People with HHT will identify themselves within the questionnaire, first by statement of what they think is their diagnosis, and second by provision of the HHT diagnostic criteria within specific questions.
  They will be directed to appropriate questions, according to answers to the previous questions.
  Interventions: Other: Questionnaire
- Controls without HHT (Other): People without HHT will identify themselves within the questionnaire, first by statement of what they think is their diagnosis, and second by provision of the HHT diagnostic criteria within specific questions.
  They will be directed to appropriate questions, according to answers to the previous questions.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — To capture large sufficiently large numbers of individuals for appropriate statistical power (see below), a web based questionnaire design was considered the most appropriate tool. SurveyMonkey was identified as the most suitable means to generate the questionnaire, facilitate confidential answers by the target populations, and for analysis of questionnaire data. The designed survey can also be presented in paper format, and used in our clinical service.
  Other Names: Survey; Confidential; SurveyMonkey SSL encryption feature; Web-link collector does not collect IP addresses

SUMMARY:
Hereditary Hemorrhagic Telangiectasia (HHT) affects 1 in 5,000 people. The purpose of this study is to provide data regarding the frequency of common health conditions and the tolerability of therapies in HHT by using a questionnaire.

This will be filled in by both people with HHT, and controls who will be members of the general population without HHT.

The questionnaire has been designed primarily for web based entry, but can also be circulated in paper format on request

DETAILED DESCRIPTION:
Hereditary Hemorrhagic Telangiectasia (HHT) affects 1 in 5,000 people, usually causing nosebleeds, skin blood spots, and/or anemia as a result of bleeding from the nose or gut. The majority of people with HHT also have abnormal blood vessels (arteriovenous malformations) in internal organs such as the lungs, liver and brain. Management of this multisystem disorder is highly challenging.

The Lead Applicant has spent 20 years working on this rare disease, and identified multiple areas where more evidence is required to assist clinicians and patients with this lifelong condition. A particular issue is what happens when people with HHT have other common medical conditions such as asthma, cancer, diabetes, or heart disease. Do they have the same pattern of problems as the general population? Can they use the same drugs? Are further safeguards needed? For these important questions, current advice can only be based on theoretical considerations and anecdotal data.

The ultimate goal of this study is to use information derived from a questionnaire to provide evidence to assist clinicians treating people with HHT.

Data will be entered from April 2012. Data will be analysed on average 6-8 months after entry.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over.
* Capacity to fill in a questionnaire.

Exclusion Criteria:

* Age under 18
* Unable to fill in a questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2174 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of nosebleeds. | Day 1
  The data outcome will be captured at the time of reporting by study participants, indicating the % of respondents affected by nosebleeds at that time. Subsequent calculations will standardise for age and other participant variables.

SECONDARY OUTCOMES:
Efficacy of nosebleed treatments | Day 1
  The data outcome will be captured at the time of reporting by study participants, indicating the % of respondents reporting beneficial, null or detrimental effects from nosebleed treatments. Subsequent calculations will standardise for age and other participant variables.

CONTACTS AND LOCATIONS:
Overall Officials: Claire L Shovlin, PhD MB BChir FRCP, Principal Investigator — Imperial College London
Locations (1):
- NHLI Cardiovascular Sciences, Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Silva BM, Hosman AE, Devlin HL, Shovlin CL. Lifestyle and dietary influences on nosebleed severity in hereditary hemorrhagic telangiectasia. Laryngoscope. 2013 May;123(5):1092-9. doi: 10.1002/lary.23893. Epub 2013 Feb 12. PMID 23404156
- [Result] Devlin HL, Hosman AE, Shovlin CL. Antiplatelet and anticoagulant agents in hereditary hemorrhagic telangiectasia. N Engl J Med. 2013 Feb 28;368(9):876-8. doi: 10.1056/NEJMc1213554. No abstract available. PMID 23445111
- [Result] Finnamore H, Le Couteur J, Hickson M, Busbridge M, Whelan K, Shovlin CL. Hemorrhage-adjusted iron requirements, hematinics and hepcidin define hereditary hemorrhagic telangiectasia as a model of hemorrhagic iron deficiency. PLoS One. 2013 Oct 16;8(10):e76516. doi: 10.1371/journal.pone.0076516. eCollection 2013. PMID 24146883
- [Result] Hosman AE, Devlin HL, Silva BM, Shovlin CL. Specific cancer rates may differ in patients with hereditary haemorrhagic telangiectasia compared to controls. Orphanet J Rare Dis. 2013 Dec 20;8:195. doi: 10.1186/1750-1172-8-195. PMID 24354965
- [Result] Elphick A, Shovlin CL. Relationships between epistaxis, migraines, and triggers in hereditary hemorrhagic telangiectasia. Laryngoscope. 2014 Jul;124(7):1521-8. doi: 10.1002/lary.24526. Epub 2014 Jan 23. PMID 24458873
- [Result] Shovlin CL, Awan I, Cahilog Z, Abdulla FN, Guttmacher AE. Reported cardiac phenotypes in hereditary hemorrhagic telangiectasia emphasize burdens from arrhythmias, anemia and its treatments, but suggest reduced rates of myocardial infarction. Int J Cardiol. 2016 Jul 15;215:179-85. doi: 10.1016/j.ijcard.2016.04.006. Epub 2016 Apr 7. PMID 27116331
- [Result] Patel T, Elphick A, Jackson JE, Shovlin CL. Injections of Intravenous Contrast for Computerized Tomography Scans Precipitate Migraines in Hereditary Hemorrhagic Telangiectasia Subjects at Risk of Paradoxical Emboli: Implications for Right-to-Left Shunt Risks. Headache. 2016 Nov;56(10):1659-1663. doi: 10.1111/head.12963. Epub 2016 Oct 11. PMID 27727478
- [Result] Shovlin CL, Patel T, Jackson JE. Embolisation of PAVMs reported to improve nosebleeds by a subgroup of patients with hereditary haemorrhagic telangiectasia. ERJ Open Res. 2016 Apr 29;2(2):00035-2016. doi: 10.1183/23120541.00035-2016. eCollection 2016 Apr. PMID 27730189
- [Result] Shovlin CL, Gilson C, Busbridge M, Patel D, Shi C, Dina R, Abdulla FN, Awan I. Can Iron Treatments Aggravate Epistaxis in Some Patients With Hereditary Hemorrhagic Telangiectasia? Laryngoscope. 2016 Nov;126(11):2468-2474. doi: 10.1002/lary.25959. Epub 2016 Apr 23. PMID 27107394
- [Result] Hosman AE, Shovlin CL. Cancer and hereditary haemorrhagic telangiectasia. J Cancer Res Clin Oncol. 2017 Feb;143(2):369-370. doi: 10.1007/s00432-016-2298-x. Epub 2016 Nov 11. PMID 27837281